CLINICAL TRIAL: NCT00241267
Title: Bronchial Ultrasonography Via a Fibrescope: Pilot Study in Tumoral Disease
Status: Terminated | Type: Observational
Sponsor: University Hospital, Tours (Other)
Other Study IDs: CT04-FT/ENDO
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2006-10-06 (Estimated); Status verified 2006-05

CONDITIONS: Pulmonary Neoplasms
Keywords: Pulmonary; Neoplasms; Endobronchial; Ultrasonography; Primary
MeSH Terms: conditions — Lung Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Device: Dedicated ultrasonographic probe during bronchoscopy

SUMMARY:
The exploration of neoplastic pulmonary pathology is based on computed tomography and bronchoscopy. This allows targeted samples of the identified lesions.

A new ultrasonographic method is proposed as a non invasive and non irradiating technic by using a dedicated probe easily introduced via the channel of the fibrescope, so as to complete the identification of peripheral lesions.

DETAILED DESCRIPTION:
The main objective of the study is to assess the ability of endobronchial ultrasonography to diagnose peripheral pulmonary lesions during the bronchoscopy and to correlate the abnormalities to computed tomography and/or histology.

The dedicated probe consist of a linear array of 2-3 mm in diameter connected to a commercial unit.

ELIGIBILITY:
Inclusion Criteria:

* Assumed proximal neoplastic pulmonary pathology
* Planned bronchoscopy and biopsy

Exclusion Criteria:

* Pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-03; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: François TRANQUART, PR, Principal Investigator — Centre d'Innovation Technologique
Locations (1):
- University Hospital of TOURS, Tours, France

REFERENCES:
- [Background] Kurimoto N, Miyazawa T, Okimasa S, Maeda A, Oiwa H, Miyazu Y, Murayama M. Endobronchial ultrasonography using a guide sheath increases the ability to diagnose peripheral pulmonary lesions endoscopically. Chest. 2004 Sep;126(3):959-65. doi: 10.1378/chest.126.3.959. PMID 15364779
- [Result] Baba M, Sekine Y, Suzuki M, Yoshida S, Shibuya K, Iizasa T, Saitoh Y, Onuma EK, Ohwada H, Fujisawa T. Correlation between endobronchial ultrasonography (EBUS) images and histologic findings in normal and tumor-invaded bronchial wall. Lung Cancer. 2002 Jan;35(1):65-71. doi: 10.1016/s0169-5002(01)00284-7. PMID 11750715
- [Result] Falcone F, Fois F, Grosso D. Endobronchial ultrasound. Respiration. 2003 Mar-Apr;70(2):179-94. doi: 10.1159/000070066. PMID 12740516